CLINICAL TRIAL: NCT05962502
Title: A Single-arm, Open-label, Phase II Clinical Study of Cetuximab Plus Irinotecan in Patients With NeoRAS Wild-type Metastatic Colorectal Cancer In Third-line Therapy
Brief Title: Cetuximab Plus Irinotecan in Patients With NeoRAS Wild-type Metastatic Colorectal Cancer In Third-line Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rui-hua Xu, MD, PhD, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEORAS-SYSUCC
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: NeoRAS wild-type; mCRC; Cetuximab; Third-line therapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cetuximab plus irinotecan (Experimental): Cetuximab 500 mg/m2 iv drip 90 min d1, Irinotecan 180 mg/m2 iv drip d1 (For patients with UGT*28 7/7 or UGT*6 A/A or UGT*28 6/7 plus UGT*6 A/G, irinotecan 150 mg/m2 is used) The above regimen is repeated every 2 weeks
  Interventions: Drug: Cetuximab and irinotecan

INTERVENTIONS:
Drug: Cetuximab and irinotecan — chemotherapy plus targeted therapy
  Other Names: ERBITUX

SUMMARY:
This is a single-arm, open-label, phase II clinical trial. The goal of this study is to evaluate the efficacy and safety of cetuximab plus irinotecan in patients with NeoRAS wild-type primary left-sided mCRC in third-line therapy.

DETAILED DESCRIPTION:
At present, the third-line therapy in China includes 3 anti-angiogenic small molecule tyrosine kinase (TKI) inhibitors, namely regorafenib, fruquintinib and oral chemotherapeutic agent TAS-102.There are high-level evidences for the above 3 drugs, but their therapeutic effects are still unsatisfactory with the progression-free survival (PFS) of only 2-4 months. As a result, more effective regimens need to be explored. The BOND study found that in mCRC patients with RAS wild-type and irinotecan resistance, cetuximab combined with irinotecan as the third-line therapy could effectively reverse irinotecan resistance with an ORR of 22.9%. The CRIKET study assessed the effect of cetuximab combined with irinotecan in later-line setting for advanced CRC; the result showed that the cetuximab combined with irinotecan therapy achieved an objective response rate (ORR) of 21% (95% CI, 10-40%). In the subgroup analysis, compared with patients with mutations, patients with RAS wild-type confirmed by circulating tumor DNA (ctDNA) had longer PFS benefit (4.0 months vs 1.9 months), which suggested that patients with RAS wild-type mCRC might still benefit from cetuximab plus irinotecan re-challenge in third-line setting after cetuximab treatment. However, third-line therapy options are still limited for another 35% to 40% patients with RAS wide-type mCRC and the prognosis for these patients is relatively poor. More studies are needed to explore other effective regimens.

ctDNA, or liquid biopsy technology, can detect DNA released from tumor cells into the blood. Moreover, it has some detecting advantages, such as real-time, dynamic, comprehensive and noninvasive. More and more studies have shown that this technology is promising and can be widely applied in the whole disease management course of CRC patients, such as early diagnosis, therapeutic target detection, minimal residual disease (MRD) detection and efficacy monitoring. One of previous studies of our team found that the status of RAS and BRAF genes detected by ctDNA in advanced CRC patients would change along with treatment. The study dynamically monitored ctDNA in 171 patients with unresectable mCRC. The results showed that 42.6% of patients with initial RAS mutation were converted to RAS wild-type mCRC after the standard first-line treatment, and such patients were called NeoRAS wild-type mCRC patients. Other studies have also found similar phenomena, but the frequency of NeoRAS wild-type conversion varies among studies (2%-45%), which might be related to several factors such as patients' treatment stage, early treatment regimen, and ctDNA detection method. Therefore, in order to optimize treatment strategies, RAS status should be retested during overall management of patients with RAS mutant mCRC.

The target population for this study is patients with RAS/BRAF wild-type primary left-sided mCRC by blood-based ctDNA testing before third-line therapy, who are initial RAS mutant and BRAF wild-type CRC patients, who have disease progression after first- and second-line therapy (previously treated with fluorouracil compounds, oxaliplatin and irinotecan) and who have tumor progression, during or within 3 months after irinotecan-containing regimen. This population will receive third-line therapy with cetuximab plus irinotecan bi-weekly until disease progression. The primary study endpoint is ORR, and the secondary study endpoints are PFS, OS and drug safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histologically confirmed colorectal adenocarcinoma.
3. Patients with initial RAS mutant, BRAF wild-type left-sided mCRC.
4. Progression after standard first-line and second-line therapy (previously treated with fluorouracil compounds, oxaliplatin and irinotecan).
5. Tumor progression within 3 months during or after irinotecan-containing regimen.
6. Blood-based ctDNA testing shows that both RAS and BRAF genes are wild-type after second-line therapy progression .
7. There are objectively measurable lesions according to RECIST v1.1 criteria.
8. Normal hematologic function (platelets > 90 × 109/L; leukocytes > 3 × 109/L; neutrophils > 1.5 × 109/L; hemoglobin > 8.0g/100ml).
9. Serum bilirubin ≤ 1.5 x the upper limit of normal (ULN) and transaminases ≤ 5 x ULN.
10. Normal coagulation function, albumin ≥ 35 g/L.
11. Liver function: Child-Push score: Class A.
12. Serum creatinine < 1.5 x ULN, or calculated creatinine clearance ≥ 50 ml/min (using the Cockcroft Gault formula).
13. ECOG PS score 0-2.
14. Life expectancy > 3 months.
15. Sign written informed consent.
16. Willing and able to be followed up until death or end of study or study termination.

Exclusion Criteria:

1. Primary right-sided mCRC.
2. dMMR/MSI-H mCRC.
3. Patients with initial RAS wild-type or BRAF mutant mCRC.
4. ctDNA testing shows that RAS or BRAF gene is mutant mCRC after second-line therapy.
5. Serious arterial embolism or ascites.
6. Serious bleeding tendency or coagulation disorder.
7. Serious uncontrolled systemic complications such as infection or diabetes.
8. Clinically significant cardiovascular disease such as cerebrovascular accident (within 6 months prior to enrollment), myocardial infarction (within 6 months prior to enrollment), uncontrolled hypertension despite appropriate medical treatment. Unstable angina, congestive heart failure (NYHA class 2-4), cardiac arrhythmia requiring medication.
9. History or physical evidence of central nervous system disease (e.g., primary brain tumor, epilepsy uncontrolled by standard of care, any history of brain metastases or stroke).
10. Other malignancies (except cutaneous basal cell carcinoma and/or cervical carcinoma in situ of the cervix and/or thyroid carcinoma after radical surgery) within the past 5 years.
11. Hypersensitivity to any drug in the study.
12. Pregnant and lactating women.
13. Women of childbearing age (< 2 years after last menstruation) or men of fertile potential who are not using or refuse to use effective non-hormonal contraception (intrauterine contraceptive ring, barrier contraceptives combined with spermicidal gel, or surgical sterilization).
14. Unable or unwilling to comply with the study protocol.
15. Patients with any other diseases, dysfunction caused by metastatic lesions, or suspected disease found by physical examination, indicating possible contraindications to the use of the investigational drug or putting the patients at high risk of treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 1 year
  Based on RECIST 1.1

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 2 years
  Based on RECIST 1.1
Overall survival (OS) | Up to 3 years
  Based on RECIST 1.1
Drug-related adverse reactions | Up to 3 years
  Based on NCI-CTCAE v5.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer center of Sun Yat-sen University, Guangzhou, Guangdong, China